CLINICAL TRIAL: NCT01054599
Title: Does Memantine Improve Verbal Memory Task Performance in Subjects With Localization-related Epilepsy and Memory Dysfunction? A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Does Memantine Improve Verbal Memory Task Performance in Subjects With Partial Epilepsy and Memory Dysfunction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Academy of Neurology (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Beth Leeman, M.D., Assistant in Neuroscience, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008P000107
Record Dates: First submitted 2009-12-01; First posted 2010-01-22 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Epilepsy
Keywords: epilepsy; memory; memantine; localization related epilepsy; focal epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — Memantine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental): Subjects will randomly assigned to take either a placebo or memantine for 13 weeks. The assignment will be double-blind, neither the study members nor the subject will know if he/she is taking memantine or a placebo.
  Interventions: Drug: Memantine
- Sugar Pill (Placebo Comparator): Subjects will be randomly assigned to take either memantine or a placebo. The study is double-blind, and neither the study members nor the subject will know if he/she is taking memantine or a placebo.
  Interventions: Other: Sugar Pill

INTERVENTIONS:
Drug: Memantine — All subjects in the treatment group will be placed on memantine. The dosage of memantine will begin at 5mg once per day (qday), and increase by 5mg every week. The titration will continue over a period of 3 weeks until a goal of 10mg bid is reached. The dosing will increase slowly, to minimize the risk of side effects. The subject will then remain on memantine at 10mg bid for 10 weeks, until the conclusion of the first phase of the study. At the conclusion of the first 13 weeks, subjects will discontinue the treatment (memantine or placebo) and enter the open label phase.
  Other Names: Namenda
  Arms: Memantine
Other: Sugar Pill — In the control arm of the study, subjects will take one placebo sugar pill per day for one week, then increase to one tablet twice per day for the following 12 weeks. At the end of this phase of the study, subjects will enter the open-label phase (unblinded treatment with memantine).
  Other Names: Placebo
  Arms: Sugar Pill
Drug: Memantine — Open label: When the blinded phase is complete (Weeks 1-13), all subjects will receive open-label treatment with memantine (Weeks 14-26). The dosage of memantine will begin at 5mg once per day (qday), and increase by 5mg every week. The titration will continue over a period of 3 weeks until a goal of 10mg bid is reached. The dosing will increase slowly, to minimize the risk of side effects. The subject will then remain on memantine at 10mg bid for 10 weeks, until the conclusion of the study. At the conclusion of the study, subjects will discontinue the treatment.
  Other Names: Namenda
  Arms: Memantine

SUMMARY:
Many patients with epilepsy have memory deficits in the setting of otherwise normal intelligence. Unfortunately, the treatment options for memory dysfunction in patients with epilepsy are limited. The investigators are conducting a study to evaluate the effects of memantine for the treatment of verbal memory dysfunction in subjects with localization-related seizures. The study involves randomization to memantine therapy or placebo, with cognitive testing and EEG pre- and post-treatment, as well as after an open-label memantine treatment phase.

The primary aim of this study is to evaluate the efficacy of memantine for the treatment of verbal memory dysfunction in subjects with left temporal lobe epilepsy. The investigators expect that verbal memory task performance will improve in those taking memantine, but not in those taking a placebo.

The investigators propose that the expected benefit of memantine is specific to verbal memory in subjects with left temporal lobe seizures, rather than representing an overall improvement in cognitive function. The investigators expect no improvement on other cognitive tasks in either the memantine or placebo groups.

The investigators will evaluate whether subjects with left temporal lobe epilepsy and memory difficulties have self-reported improvement in memory while taking memantine. The investigators expect improvement of self-rated memory function on the Quality of Life in Epilepsy Patient Inventory (QOLIE-89) in the memantine group, but no change on this scale in the placebo group.

DETAILED DESCRIPTION:
Patients with epilepsy frequently demonstrate subtle cognitive difficulties in the setting of otherwise normal intelligence. Those with left temporal lobe seizures often have particular deficits in verbal memory (Blum 2001). These memory difficulties may be the most distressing aspect of epilepsy for the patients.

Unfortunately, treatment options for memory dysfunction are limited. Cognitive therapy, for example, may help patients to cope, but does not treat the memory loss or address the underlying pathologic process. Two studies examined the pharmacologic management of memory dysfunction in patients with epilepsy using donepezil (Aricept), but with inconsistent results and questionable benefit. A pilot study by Fisher et al. (2001) showed some promise for use of the drug. The study found improved immediate recall and consistent long-term retrieval scores on the Buschke Selective Reminding Test after three months of open-label treatment when compared to a pre-treatment baseline. A more recent randomized, double-blind, placebo-controlled cross-over trial of donepezil, however, showed no effect on memory as measured by delayed recall on the Hopkins Verbal Learning Test (Hamberger et al. 2007).

Use of donepezil, an acetylcholinesterase inhibitor, may pose a risk of seizure exacerbation in this population. Fisher et al. (2001) reported a significant increase in the frequency of generalized tonic-clonic seizures during donepezil treatment. Cholinergic agents have been shown to cause seizures in animal models as well (Turski et al. 1989). Given isolated case reports of seizures associated with donepezil use, the manufacturer issued an advisory note warning of a possible relationship, although data have been insufficient to establish causality. While an increase in seizures was not noted in the Hamberger et al. (2007) study, seizure exacerbation remains a concern regarding the use of this drug in patients with epilepsy.

The mechanism for the postulated effect of donepezil is unclear. Cholinergic transmission has not traditionally been viewed as a contributor to hippocampal pathology. It is believed that excitotoxicity, mediated by glutamate acting on NMDA receptors in the hippocampus, causes hippocampal sclerosis. This process leads to further seizures and memory dysfunction. Alteration of this excitotoxic pathway would be a novel, and potentially safer and more effective, approach to the treatment of memory loss.

The possible effect of intervention at the level of excitotoxicity is supported by animal data. Such studies demonstrate that induced seizures in a rat model of epilepsy will lead to decrements in performance of a spatial memory task, the Morris water maze. This memory dysfunction, however, can be mitigated by NMDA antagonists, such as MK-801, administered prior to seizure induction. The underlying concept is that NMDA receptor antagonists would block the pathway of excitotoxicity that leads to hippocampal injury and memory loss (Kelsey et al. 2000).

An NMDA antagonist, memantine (Namenda), is prescribed in humans for treatment of moderate to severe Alzheimer's disease (Tariot et al. 2004, Reisberg et al. 2003, 2006). Patients with Alzheimer's disease have attained significant cognitive improvements with use of the drug, as measured by the Severe Impairment Battery. The time-course of benefit is less clear, with some studies demonstrating sustained improvement (Tariot et al. 2004) and others showing more transient benefits over the first several weeks of treatment (Reisberg et al. 2003).

It is unknown, however, if an NMDA antagonist such as memantine would be of benefit in humans with memory dysfunction and seizures. The proposed study tests the hypothesis that treatment with memantine would improve verbal memory test performance in patients with localization-related epilepsy. If beneficial, this would provide a much-needed treatment option.

The study will examine the primary specific aim:

Aim 1: Improvement in memory test performance. The primary aim of this study is to evaluate the efficacy of memantine for the treatment of verbal memory dysfunction in subjects with left temporal lobe epilepsy. We expect that verbal memory task performance, as measured by the Buschke Selective Reminding Test (SRT), will improve in those taking memantine, but not while taking a placebo. Such a finding would support the use of memantine for treatment of memory loss in this population, as well as more generally support the hypothesis that NMDA receptor hyperactivity is an appropriate target for intervention.

The study will examine two secondary specific aims:

Aim 2: Selectivity of response. We propose that the postulated benefit of memantine is specific to verbal memory in subjects with left temporal lobe seizures, and visuospatial memory in subjects with right temporal lobe seizures, rather than representing an overall improvement in cognitive function. We expect no improvement on other cognitive tasks in either the memantine or placebo groups, with measures including the Digit Span (for sustained attention, immediate span), Spatial Span (for visuospatial working memory and span), Block Design (for visuospatial construction), Verbal Fluency, Design Fluency, and Stroop Color Word Interference (for executive function) tests. This would lend support to the hypothesis that blockade of NMDA receptor hyperactivity in the hippocampus would lead to improved performance on cognitive tasks that depend specifically on the integrity of that hippocampus, as opposed to a general benefit in overall cognition.

Aim 3: Improvement in self-reported memory function. We will evaluate whether subjects with localization-related epilepsy and memory difficulties have subjective improvement in memory with the administration of memantine. We expect improvement of self-rated memory function on the Quality of Life in Epilepsy Patient Inventory (QOLIE-89) with memantine, but no change on this scale with placebo. This measure serves to evaluate the hypothesis that memantine treatment leads to clinically meaningful improvement.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Normal IQ as estimated by the Wechsler Test of Adult Reading (WTAR)
* Able to give consent
* Able to live independently and complete activities of daily living
* Stable frequency of seizures. There is no minimum/maximum criteria for the frequency of partial seizures. Those with infrequent secondary generalized seizures may participate, with infrequent seizures defined as two or fewer per year.
* The subject's treating physician does not believe a change in anticonvulsant regimen to be warranted. The anticonvulsant drugs must remain unchanged during the 26 week trial.
* Partial-onset seizures. Seizure type will be determined by clinical history, MRI, SPECT and/or PET imaging, and interictal and/or ictal EEG.
* Either symptomatic or idiopathic seizures.

Exclusion Criteria:

* Non-epileptic seizures
* Prior surgical resection for treatment of seizures
* Progressive neurologic illness (i.e. tumor evident on MRI)
* Current alcohol or drug abuse, as this may affect memory by other mechanisms. This information may be obtained by self-report, from the referring physician or by medical record.
* Diagnosis of Alzheimer's disease, nutritional deficiency, infection or metabolic/electrolyte disorder causing memory loss.
* Non-native English speaking and/or multilingual.
* Seizure(s) must not have occurred within 3 days of testing.
* Subjects who are pregnant will not be eligible to take part in the study, as memantine is classified as a Pregnancy Category B drug and may pose risk to the fetus.
* Women who are breastfeeding may not participate in this study.
* Those with renal tubular acidosis or infections of the urinary tract will not be eligible for participation, as memantine is renally cleared and conditions that alkalinize the urine may reduce clearance of the drug.
* Subjects with severe renal impairment, defined as a creatinine clearance of ≤29 mL/min, will be excluded as such patients may not tolerate the proposed dosing schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Moo, M.D., Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts

REFERENCES:
- [Background] Blum D. Decline in Verbal Memory Associated with Duration of Epilepsy: An Intracarotid Amobarbital Study. Epilepsy Behav. 2001 Oct;2(5):448-453. doi: 10.1006/ebeh.2001.0239. PMID 12609282
- [Background] Busch RM, Frazier TW, Haggerty KA, Kubu CS. Utility of the Boston naming test in predicting ultimate side of surgery in patients with medically intractable temporal lobe epilepsy. Epilepsia. 2005 Nov;46(11):1773-9. doi: 10.1111/j.1528-1167.2005.00300.x. PMID 16302857
- [Background] Diaz-Asper CM, Dopkins S, Potolicchio SJ Jr, Caputy A. Spatial memory following temporal lobe resection. J Clin Exp Neuropsychol. 2006 Nov;28(8):1462-81. doi: 10.1080/13803390500434359. PMID 17050270
- [Background] Dodrill CB, Ojemann GA. Do recent seizures and recent changes in antiepileptic drugs impact performances on neuropsychological tests in subtle ways that might easily be missed? Epilepsia. 2007 Oct;48(10):1833-41. doi: 10.1111/j.1528-1167.2007.01140.x. Epub 2007 May 23. PMID 17521340
- [Background] Fisher RS, Bortz JJ, Blum DE, Duncan B, Burke H. A pilot study of donepezil for memory problems in epilepsy. Epilepsy Behav. 2001 Aug;2(4):330-4. doi: 10.1006/ebeh.2001.0221. PMID 12609209
- [Background] Halsband U. Bilingual and multilingual language processing. J Physiol Paris. 2006 Jun;99(4-6):355-69. doi: 10.1016/j.jphysparis.2006.03.016. Epub 2006 May 24. PMID 16723214
- [Background] Hamberger MJ, Palmese CA, Scarmeas N, Weintraub D, Choi H, Hirsch LJ. A randomized, double-blind, placebo-controlled trial of donepezil to improve memory in epilepsy. Epilepsia. 2007 Jul;48(7):1283-91. doi: 10.1111/j.1528-1167.2007.01114.x. Epub 2007 May 1. PMID 17484756
- [Background] Helmstaedter C, Elger CE, Lendt M. Postictal courses of cognitive deficits in focal epilepsies. Epilepsia. 1994 Sep-Oct;35(5):1073-8. doi: 10.1111/j.1528-1157.1994.tb02557.x. PMID 7925154
- [Background] Hermann BP, Seidenberg M, Schoenfeld J, Peterson J, Leveroni C, Wyler AR. Empirical techniques for determining the reliability, magnitude, and pattern of neuropsychological change after epilepsy surgery. Epilepsia. 1996 Oct;37(10):942-50. doi: 10.1111/j.1528-1157.1996.tb00531.x. PMID 8822692
- [Background] Kelsey JE, Sanderson KL, Frye CA. Perforant path stimulation in rats produces seizures, loss of hippocampal neurons, and a deficit in spatial mapping which are reduced by prior MK-801. Behav Brain Res. 2000 Jan;107(1-2):59-69. doi: 10.1016/s0166-4328(99)00107-2. PMID 10628730
- [Background] Kim KH, Relkin NR, Lee KM, Hirsch J. Distinct cortical areas associated with native and second languages. Nature. 1997 Jul 10;388(6638):171-4. doi: 10.1038/40623. PMID 9217156
- [Background] Lee S, Sziklas V, Andermann F, Farnham S, Risse G, Gustafson M, Gates J, Penovich P, Al-Asmi A, Dubeau F, Jones-Gotman M. The effects of adjunctive topiramate on cognitive function in patients with epilepsy. Epilepsia. 2003 Mar;44(3):339-47. doi: 10.1046/j.1528-1157.2003.27402.x. PMID 12614389
- [Background] Lucas TH 2nd, McKhann GM 2nd, Ojemann GA. Functional separation of languages in the bilingual brain: a comparison of electrical stimulation language mapping in 25 bilingual patients and 117 monolingual control patients. J Neurosurg. 2004 Sep;101(3):449-57. doi: 10.3171/jns.2004.101.3.0449. PMID 15352603
- [Background] Lutz MT, Helmstaedter C. EpiTrack: tracking cognitive side effects of medication on attention and executive functions in patients with epilepsy. Epilepsy Behav. 2005 Dec;7(4):708-14. doi: 10.1016/j.yebeh.2005.08.015. Epub 2005 Nov 2. PMID 16266826
- [Background] McLean MJ, Gupta RC, Dettbarn WD, Wamil AW. Prophylactic and therapeutic efficacy of memantine against seizures produced by soman in the rat. Toxicol Appl Pharmacol. 1992 Jan;112(1):95-103. doi: 10.1016/0041-008x(92)90284-y. PMID 1733053
- [Background] Meador KJ, Loring DW, Vahle VJ, Ray PG, Werz MA, Fessler AJ, Ogrocki P, Schoenberg MR, Miller JM, Kustra RP. Cognitive and behavioral effects of lamotrigine and topiramate in healthy volunteers. Neurology. 2005 Jun 28;64(12):2108-14. doi: 10.1212/01.WNL.0000165994.46777.BE. PMID 15985582
- [Background] Reisberg B, Doody R, Stoffler A, Schmitt F, Ferris S, Mobius HJ; Memantine Study Group. Memantine in moderate-to-severe Alzheimer's disease. N Engl J Med. 2003 Apr 3;348(14):1333-41. doi: 10.1056/NEJMoa013128. PMID 12672860
- [Background] Reisberg B, Doody R, Stoffler A, Schmitt F, Ferris S, Mobius HJ. A 24-week open-label extension study of memantine in moderate to severe Alzheimer disease. Arch Neurol. 2006 Jan;63(1):49-54. doi: 10.1001/archneur.63.1.49. PMID 16401736
- [Background] Sabsevitz DS, Swanson SJ, Morris GL, Mueller WM, Seidenberg M. Memory outcome after left anterior temporal lobectomy in patients with expected and reversed Wada memory asymmetry scores. Epilepsia. 2001 Nov;42(11):1408-15. doi: 10.1046/j.1528-1157.2001.38500.x. PMID 11879343
- [Background] Schefft BK, Testa SM, Dulay MF, Privitera MD, Yeh HS. Preoperative assessment of confrontation naming ability and interictal paraphasia production in unilateral temporal lobe epilepsy. Epilepsy Behav. 2003 Apr;4(2):161-8. doi: 10.1016/s1525-5050(03)00026-x. PMID 12697141
- [Background] Stroup E, Langfitt J, Berg M, McDermott M, Pilcher W, Como P. Predicting verbal memory decline following anterior temporal lobectomy (ATL). Neurology. 2003 Apr 22;60(8):1266-73. doi: 10.1212/01.wnl.0000058765.33878.0d. PMID 12707428
- [Background] Tariot PN, Farlow MR, Grossberg GT, Graham SM, McDonald S, Gergel I; Memantine Study Group. Memantine treatment in patients with moderate to severe Alzheimer disease already receiving donepezil: a randomized controlled trial. JAMA. 2004 Jan 21;291(3):317-24. doi: 10.1001/jama.291.3.317. PMID 14734594
- [Background] Turski L, Ikonomidou C, Turski WA, Bortolotto ZA, Cavalheiro EA. Review: cholinergic mechanisms and epileptogenesis. The seizures induced by pilocarpine: a novel experimental model of intractable epilepsy. Synapse. 1989;3(2):154-71. doi: 10.1002/syn.890030207. PMID 2648633
- [Background] Zipf-Williams EM, Shear PK, Strongin D, Winegarden BJ, Morrell MJ. Qualitative block design performance in epilepsy patients. Arch Clin Neuropsychol. 2000 Feb;15(2):149-57. PMID 14590558
- [Derived] Leeman-Markowski BA, Meador KJ, Moo LR, Cole AJ, Hoch DB, Garcia E, Schachter SC. Does memantine improve memory in subjects with focal-onset epilepsy and memory dysfunction? A randomized, double-blind, placebo-controlled trial. Epilepsy Behav. 2018 Nov;88:315-324. doi: 10.1016/j.yebeh.2018.06.047. Epub 2018 Oct 27. PMID 30449328

RESULTS

PARTICIPANT FLOW:
Groups:
- Memantine: Subjects will randomly assigned to take either a placebo or memantine for 13 weeks. The assignment will be double-blind, neither the study members nor the subject will know if he/she is taking memantine or a placebo.
  Memantine: The dosage of memantine will begin at 5mg once per day (qday), and increase by 5mg every week. The titration will continue over a period of 3 weeks until a goal of 10mg bid is reached. The subject will then remain on memantine at 10mg bid for 10 weeks, until the conclusion of the first phase of the study. At the conclusion of the first 13 weeks, subjects will discontinue the treatment (memantine or placebo) and enter the open label phase.
- Sugar Pill: Subjects will be randomly assigned to take either memantine or a placebo. The study is double-blind, and neither the study members nor the subject will know if he/she is taking memantine or a placebo.
  Sugar Pill: In the control arm of the study, subjects will take one placebo sugar pill per day for one week, then increase to one tablet twice per day for the following 12 weeks. At the end of this phase of the study, subjects will enter the open-label phase (unblinded treatment with memantine). The dosage of memantine will begin at 5mg once per day (qday), and increase by 5mg every week. The titration will continue over a period of 3 weeks until a goal of 10mg bid is reached. The subject will then remain on memantine at 10mg bid for 10 weeks, until the conclusion of the study
Period: Overall Study
Arm/Group | Memantine | Sugar Pill
Started | 13 | 16
Completed | 9 | 9
Not Completed | 4 | 7
Not completed — Dizziness due to phenytoin toxicity | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Spells/seizure-like episodes | 1 | 1
Not completed — Timing/scheduling difficulties | 1 | 1
Not completed — Visual impairment, WTAR <80 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Sugar Pill | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (13.1) | 45.3 (12.6) | 44.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/Caucasian | 11 | 16 | 27
  Race/Ethnicity: Black or African American | 1 | 0 | 1
  Race/Ethnicity: Hispanic or Latino | 1 | 0 | 1
  Race/Ethnicity: American Indian or Alaska Native | 0 | 0 | 0
  Race/Ethnicity: Asian | 0 | 0 | 0
  Race/Ethnicity: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race/Ethnicity: Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Change Scores in Memory Measures From Baseline to Post-treatment/Placebo Will be Compared Between the Memantine Treatment and Placebo Groups.
Description: Change scores from pre- to post-treatment/placebo were calculated for the primary outcome measures, the Selective Reminding Test Continuous Long-Term Retrieval (range 0-72; higher scores indicate better memory) and 7-24 Spatial Recall Test Total Learning (range 0-35; total correct across 5 learning trials are summed, with higher scores indicating better memory) scores. These measures are scores on a scale, rather than representing standard units.
Time Frame: 13 weeks
Population: The analysis includes subjects who completed both sessions 1 (baseline) and 2 (post-treatment/placebo). One subject in the memantine group completed both sessions, but the data were excluded from analysis due to seizures occurring during testing sessions 1 and 2, yielding n=8 in the memantine group.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Memantine | Sugar Pill
Number analyzed (Participants) | 8 | 9
scores on a scale
  7-24 Spatial Recall Tests Learning Change Score | 1.00 (2.00) | 1.78 (4.99)
  SRT Continuous Long-Term Retrieval Change Score | 4.38 (7.6) | 8.11 (9.51)
Statistical Analysis 1: Comparison: Memantine vs Sugar Pill; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: To Test the Hypothesis That Improvement Will be Selective for Verbal Memory, Change Scores on the Non-verbal Tasks Will be Compared Between the Placebo and Memantine Treatment Groups.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2017-12

3. Secondary Outcome: To Test the Hypothesis That Treatment With Memantine Will Result in Subjective Improvement of Memory Function, the Change Scores From the QOLIE-89 Will be Evaluated.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2017-12

4. Secondary Outcome: A Secondary Analysis Will Examine the Possible Sustained Benefit of Continued Memantine Use.
Description: SRT-CLTR (range 0-72; higher scores indicate better memory), and 7-24 Spatial Memory Test (range 0-35; scores are summed across the 5 learning trials, with higher scores indicating better memory) scores will be assessed across the first (baseline) and third (post-open label memantine) testing sessions. These measures are considered to be scores on a scale, rather than standard units. The hypothesis was that subjects randomized to memantine would demonstrate sustained improvement from baseline, while the placebo group would demonstrate improvements after taking open label memantine (compared to baseline).
Time Frame: 26 weeks
Population: This analysis included only those subjects who participated in the open label extension period.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Memantine | Sugar Pill
Number analyzed (Participants) | 3 | 7
scores on a scale
  SRT CLTR Baseline | 32.67 (14.01) | 22.71 (9.09)
  SRT CLTR Post-Open Label | 40.33 (16.77) | 40.29 (18.81)
  7-24 Total Learning Baseline | 30.33 (4.04) | 28.14 (5.67)
  7-24 Total Learning Post-Open Label | 31.67 (4.93) | 32.43 (2.94)
Statistical Analysis 1: Comparison: Memantine vs Sugar Pill; Test type: Other; p > 0.05, Wilcoxon Signed Ranks Test

ADVERSE EVENTS:
Arm/Group | Memantine | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/13 | 2/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=13) | Sugar Pill (N=16)
Dizziness (due to phenytoin toxicity) (Nervous system disorders) | 1 (1) | 0 (0)
Increase/recurrence of seizure-like episodes (Nervous system disorders) | 1 (1) | 1 (1)
Generalized convulsion/seizure (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No